CLINICAL TRIAL: NCT00946738
Title: A Prospective Randomized Controlled Study Analyzing the Effect of Biofeedback and Deep Oscillation on Raynaud´s Phenomenon Secondary to Systemic Sclerosis
Brief Title: The Effect of Physical Therapy on Raynaud's Phenomenon Secondary to Systemic Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Physiomed Elektromedizin AG Germany (Unknown)
Responsible Party: Anett Reißhauer MD, Department of Physical Medicine and Rehabilitation , Charité Berlin
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: EA 1/100/05
Record Dates: First submitted 2009-07-24; First posted 2009-07-27 (Estimated); Last update posted 2009-07-27 (Estimated); Status verified 2009-07

CONDITIONS: Raynaud's Phenomenon; Systemic Sclerosis
Keywords: Raynaud's phenomenon; biofeedback; deep oscillation; systemic sclerosis; physiotherapy
MeSH Terms: conditions — Raynaud Disease; Scleroderma, Systemic | interventions — Biofeedback, Psychology

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- physical therapy (Active Comparator)
  Interventions: Other: Biofeedback; Other: Deep oscillation
- control (No Intervention)

INTERVENTIONS:
Other: Biofeedback — Biofeedback training as behaviour treatment was performed thrice weekly for 4 week.
  Arms: physical therapy
Other: Deep oscillation — Deep oscillation providing a pulsing electromagnetic field was performed thrice weekly for 4 weeks.
  Arms: physical therapy

SUMMARY:
The effect of deep oscillation and biofeedback on Raynaud's phenomenon secondary to systemic sclerosis (SSc) remains to be determined. A prospective randomized controlled pilot study was performed in SSc patients receiving either deep oscillation, biofeedback thrice a week for four weeks or were randomized to the control group.

ELIGIBILITY:
Inclusion Criteria:

* ACR criteria for SSc

Exclusion Criteria:

* acute inflammatory disease, Valentini Score>3

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28
Dates: Start 2004-10; Primary Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
RP score , measured by a visual analogue scale (VAS) | 12 weeks

SECONDARY OUTCOMES:
ulceration of the skin and general disease symptoms using analogous VAS-scores | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physical Medicine and Rehabilitation , Charité University Hospital Berlin, Berlin, 10117, Germany

REFERENCES:
- [Derived] Sporbeck B, Mathiske-Schmidt K, Jahr S, Huscher D, Becker M, Riemekasten G, Taufmann I, Burmester GR, Pogel S, Reisshauer A. Effect of biofeedback and deep oscillation on Raynaud's phenomenon secondary to systemic sclerosis: results of a controlled prospective randomized clinical trial. Rheumatol Int. 2012 May;32(5):1469-73. doi: 10.1007/s00296-011-1882-2. Epub 2011 Apr 8. PMID 21476099